CLINICAL TRIAL: NCT02035527
Title: A Phase I/II Clinical Trial of Sorafenib in Combination With Cisplatin and Docetaxel in Patients With Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Sorafenib Tosylate, Cisplatin, and Docetaxel in Treating Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Matthew Old, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-13141; NCI-2013-02086 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Salivary Gland Squamous Cell Carcinoma; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IVA Salivary Gland Cancer; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Oral Cavity Squamous Cell Carcinoma; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Salivary Gland Cancer; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Salivary Gland Cancer; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Verrucous Carcinoma of the Larynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer; Untreated Metastatic Squamous Neck Cancer With Occult Primary
Keywords: squamous cell carcinoma; head and neck
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms; Carcinoma, Squamous Cell | interventions — Sorafenib; Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sorafenib tosylate, docetaxel, and cisplatin) (Experimental): Patients receive sorafenib tosylate PO BID on days 1-14 of course 0. Beginning in course 1, patients receive sorafenib tosylate PO BID on days 1-21, docetaxel IV over 1 hour on day 1, and cisplatin IV over 1 hour on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive sorafenib tosylate PO BID in the absence of disease progression or unacceptable toxicity.Correlative studies will be performed and a total of three biopsies (blood and tumor samples) will be obtained in consenting patients.Pre-treatment biopsy to establish diagnosis and baseline data, Research biopsy obtained at the end of a two week period of sorafenib monotherapy just prior to administration of cycle1 with cisplatin and docetaxel, Research biopsy obtained at the end of two chemotherapy cycles.
  Interventions: Drug: sorafenib tosylate; Drug: cisplatin; Drug: docetaxel; Other: Correlative Studies

INTERVENTIONS:
Drug: sorafenib tosylate — Given daily PO in the a.m.
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Drug: cisplatin — Given IV over 1 hour following Docetaxel administration
  Other Names: CACP; CDDP; CPDD; DDP
Drug: docetaxel — Given IV 1 hour prior to cisplatin administration
  Other Names: RP 56976; Taxotere; TXT
Other: Correlative Studies — Correlative studies will be performed at the following time points. A total of three biopsies (blood and tumor samples) will be obtained in consenting patients.Pre-treatment biopsy to establish diagnosis and baseline data, Research biopsy obtained at the end of a two week period of sorafenib monotherapy just prior to administration of cycle1 with cisplatin and docetaxel, Research biopsy obtained at the end of two chemotherapy cycles.
  Other Names: laboratory biomarker analysis

SUMMARY:
This phase I/II trial studies the side effects and the best dose of sorafenib tosylate and docetaxel when given together with cisplatin and to see how well they work in treating patients with recurrent or metastatic squamous cell carcinoma of the head and neck. Drugs used in chemotherapy, such as cisplatin and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sorafenib tosylate may also help cisplatin and docetaxel work better by making tumor cells more sensitive to the drugs. Giving sorafenib tosylate, cisplatin, and docetaxel may be an effective treatment for squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define progression-free survival of patients with recurrent/metastatic squamous cell carcinoma treated with cisplatin/docetaxel/sorafenib (sorafenib tosylate) (CDS) combination chemotherapy. (Phase II) II. To determine the optimal doses of cisplatin/docetaxel/sorafenib to be used in the phase II portion of the trial. (Phase I)

SECONDARY OBJECTIVES:

I. To determine overall survival, response rate, conduct biomarker studies, toxicities.

OUTLINE: This is a phase I, dose-escalation study of sorafenib tosylate and docetaxel followed by a phase II study.

Patients receive sorafenib tosylate orally (PO) twice daily (BID) on days 1-14 of course 0. Beginning in course 1, patients receive sorafenib tosylate PO BID on days 1-21, docetaxel intravenously (IV) over 1 hour on day 1, and cisplatin IV over 1 hour on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive sorafenib tosylate PO BID in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic or cytologic proof of recurrent/metastatic squamous cell carcinoma of the head and neck (SCCHN) of any primary site, including unknown primary cancers of the head and neck excluding nasopharyngeal carcinoma of histologic types World Health Organization (WHO) 2 or 3, paranasal sinuses primary or squamous cell carcinoma that originated in the skin
* Patients must have SCCHN that is either (a) recurrent, judged incurable by surgery or (chemo)radiation or (b) metastatic
* Patients must not have received prior chemotherapy for recurrent or metastatic disease
* Patients may have received one regimen of induction, concomitant chemoradiotherapy and/or adjuvant chemotherapy as part of their initial treatment with curative intent, which must have been completed for a minimum of 4 months prior to study treatment and patient must have been progression-free for at least 4 months since completion of treatment with curative intent
* Patients with recurrent disease are allowed a maximum of one prior radiation therapy regimen, either curative or palliative
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1
* Patients must have measurable disease using Response Evaluation Criteria in Solid Tumors (RECIST) criteria; patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Absolute neutrophil count (ANC) 1500/mm^3
* Platelet count 100,000/mm^3
* Creatinine within normal limits (WNL), or creatinine clearance >= 60 ml/min, based on the Cockroft-Gault formula
* Total bilirubin WNL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than twice the upper normal limit
* Patients must have controlled blood pressure (150/90) prior to initiation of treatment
* Women must not be pregnant or breast feeding; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of sorafenib administration
* Patients must be human immunodeficiency virus (HIV)-negative
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 months prior to entering the study
* Patients who are receiving any other investigational agents
* Patients with known brain metastases will be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib, docetaxel, cisplatin
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Uncontrolled hypertension (systolic pressure > 140 mm Hg or diastolic pressure > 90 mm Hg [National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0] on repeated measurement) despite optimal medical management
* Evidence or history of bleeding diathesis or coagulopathy
* Subject with any pulmonary hemorrhage/bleeding event of NCI-CTCAE v4.0 grade 2 or higher within 4 weeks before randomization; any other hemorrhage/bleeding event of NCI-CTCAE v4.0 grade 3 or higher within 4 weeks before randomization
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) within 6 months of informed consent
* Subjects who have used strong cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) inducers (e.g., phenytoin, carbamazepine, phenobarbital, St. John's Wort [Hypericum perforatum], or rifampin [rifampicin], and/or rifabutin) within 28 days before randomization
* Subjects with any previously untreated or concurrent cancer that is distinct in primary site or histology from breast cancer except cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor; subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before randomization are allowed; all cancer treatments must be completed at least 3 years prior to study entry (i.e., signature date of the informed consent form)
* History of organ allograft; (including corneal transplant)
* Any malabsorption condition
* Inability to comply with the protocol
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) as graded according to the NCI-CTCAE v4.0 (Phase I) | Day 21 of course 1
  A DLT will be considered a grade 3 non-hematologic toxicity or grade 4 hematologic toxicity that are probably or definitely related to treatment and result in treatment delay of more than 14 days.
Progression-free survival (PFS) (Phase II) | Time of enrollment to the date of progression diagnosis or death, assessed up to 4 weeks after completion of study treatment
  PFS will be estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 4 weeks after completion of study treatment
  OS will be estimated using the Kaplan-Meier method.
Response rate evaluated by RECIST v1.1 | Up to 4 weeks after completion of study treatment
Biomarker levels | Up to 42 days
  Biomarkers from tissue and blood samples will be evaluated and correlated with outcome parameters. Correlative biomarkers will be analyzed using mixed model for repeated measurement to account for the association of measures overtime from the same patient.
Incidence of toxicities, graded according to NCI-CTCAE version 4.0 | Up to 4 weeks after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Old, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu